CLINICAL TRIAL: NCT06161922
Title: Real World Patient-Reported Outcomes in Chinese Her2+ Early Breast Cancer Patients Receiving (Neo) Adjuvant Anti-Her2 Based Therapy
Brief Title: Real World Patient-Reported Outcomes in Chinese Her2+ EBC Patients Receiving (Neo) Adjuvant Anti-Her2 Based Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Keda Yu, Professor, Fudan University
Other Study IDs: ML44677
Record Dates: First submitted 2023-11-14; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: HER2-positive Breast Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a non-interventional observational, multi-center cohort study to evaluate patient-reported outcomes in Chinese HER2+ early breast cancer patients undergoing (neo) adjuvant anti-HER2 based therapy and describe changes over time, from baseline to 12 months.

DETAILED DESCRIPTION:
This is a non-interventional observational, multi-center cohort study with primary prospective data collection. This study will be conducted at approximately 10 sites in China.

The study population is Chinese HER2+ early breast cancer patients receiving (neo) adjuvant anti-HER2 based therapy.

Patients who are eligible for (neo) adjuvant anti-HER2 based therapy will enroll in this study.

Treatment choice in this non-interventional study will be at the discretion of the treating physician as per CACA-CBCS guidelines.

Participants are longitudinally assessed at baseline (T0, before treatment), during chemotherapy (T1, after 2 cycles), 1-month after completion of chemotherapy (T2) and at 12-month follow-up (T3).

The PRO instruments will be captured by electronic devices through WeChat mini-program which are input by patients, before or after their clinic visit but before administration of anti-HER2 therapy. Paper questionnaires will be available only as a last option if the electronic devices cannot be used for any reason (such as issues with internet access or if the device is not working). Oncology staff provided no assistance with filling in the questionnaires, but a prerecorded video will provide a detailed explanation of the questionnaires before the ePRO questionnaires. The PROs data will be restored centrally at the server of the leading site.

The usage of PROs is considered non-interventional according to local regulation. PRO measures include EORTC QLQ-C30, PDQ-5 (cognitive), PHQ-9 (depression), GAD-7 (anxiety) and Insomnia Severity Index (ISI).

Patient satisfaction for subcutaneous injection will be assessed using TASQ-SC at T3.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years;
2. Women;
3. Have signed the informed consent form as per local regulations;
4. Newly diagnosed with non-metastatic breast cancer (stage I-II-III, HER2+) at the time of starting anti-HER2 therapy;
5. Be able to comply with the follow-up visits, assessments, answering questionnaires.

Exclusion Criteria:

1. Metastatic breast cancer;
2. Prior systemic treatment for any malignancy;
3. Active secondary cancer requiring anti-HER2 therapy;
4. Vulnerable populations [e.g., decisional impaired (cognitive, psychiatric), terminally ill, prisoners], or patients who, in the opinion of the investigator have a condition that precludes their ability to provide an informed consent;
5. Men.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is Chinese HER2+ early breast cancer patients receiving (neo) adjuvant anti-HER2 based therapy. Patients who are eligible for (neo) adjuvant anti-HER2 based therapy will enroll in this study.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
EORTC QLQ-C30 score | Through study completion, an average of 1 year.
  EORTC QLQ C30 /+ BR23(EORTC breast cancer-specific quality of life) questionnaire to evaluate quality of life.
  Participants report the extent to which they have experienced those symptoms or problems during the past week. Each of the symptoms or problems is indicated with four extents, including "not at all" for 1 score, "a little" for 2 score, "quit a bit" for 3 score and "very much" for 4 score. A higher score indicated a worse quality of life.

SECONDARY OUTCOMES:
PDQ-5 score | Through study completion, an average of 1 year.
  Perceived Deficits Questionnaire to capture decline in cognitive function. Participants report the extent to which they have experienced those symptoms or problems during the past week. Each of the symptoms or problems is indicated with four extents, including " never" for 0 score, "rarely" for 1 score, " sometimes" for 2 score and " often" for 3 score, "almost always"for 4 score. A higher score indicated a more serious decline in cognitive function.
PHQ-9 score | Through study completion, an average of 1 year.
  Patient Health Questionnaire to measure the severity of depression. Participants report the extent to which they have experienced those symptoms or problems during the past week. Each of the symptoms or problems is indicated with four extents, including "not at all" for 0 score," several days " for 1 score, " more than half the days " for 2 score and " nearly every day " for 3 score. A higher score indicated a worse state.
GAD-7 score | Through study completion, an average of 1 year.
  GAD-7 (Generalized Anxiety Disorder-7) questionnaire to evaluate anxiety: includes scores for all 7 items and date of self-assessment at T0 to T3.
  Participants report the extent to which they have experienced those symptoms or problems during the past week. Each of the symptoms or problems is indicated with four extents, including "not at all" for 0 score," several days " for 1 score, " more than h
ISI score | Through study completion, an average of 1 year.
  ISI (Insomnia Severity Index) questionnaire to evaluate Insomnia Severity: includes scores for all 7 items and date of self-assessment .
  Participants report the extent to which they have experienced those symptoms or problems during the past two weeks. Each of the symptoms or problems is indicated with four extents, the total value range from 0 to 21, and higher scores mean a more severe insomnia.
TASQ-SC score | Through study completion, an average of 1 year.
  Therapy Administration Satisfaction Questionnaire is a 12-item questionnaire measuring the impact of each mode of treatment administration on five domains: physical impact, psychological impact, impact on activities of daily living, convenience, and satisfaction. Each of the domain/scale scores is scored on a 1-100 scale, where 0 is worst and 100 is best.

OTHER OUTCOMES:
Demographics characteristics | Through study completion, an average of 1 year.
  Demographics characteristics: include age, height in meters, weight in kilograms, and WHO Performance Status score.
  The age of the patients will be measured in years, height will be documented by meters, weight by kilograms, and WHO Performance Status score will be classified into 0-4 levels.
  0: able to carry out all normal activity without restriction.
  1. restricted in strenuous activity but ambulatory and able to carry out light work.
  2. ambulatory and capable of all self-care but unable to carry out any work activities; up and about more than 50% of waking hours.
  3. symptomatic and in a chair or in bed for greater than 50% of the day but not bedridden.
  4. completely disabled; cannot carry out any self-care; totally confined to bed or chair.
Socio-economic status | Through study completion, an average of 1 year.
  Socio-economic status: include income, education, and marital status.
Clinical characteristics | Through study completion, an average of 1 year.
  Clinical characteristics: include assessment of the primary site, histology, TNM stage, histological grade, ER/PR status, which will obtained from the pathology results.
  The primary site will be documented by surgeons and pathologists, histology will be decided by pathologists, TNM stage will be recorded according to the pathology results, histological grade will be documented by WHO grade I to III, ER/PR status will be measured with immumohistochemical staining.
Treatment sequence (neoadjuvant vs adjuvant) checklist | Through study completion, an average of 1 year.
  Patients receiving neoadjuvant or adjuvant treatments in fact.
Clinical treatment checklist | Through study completion, an average of 1 year.
  Clinical treatment: include breast surgery (Mastectomy vs Conservative surgery), axillary surgery (axillary dissection vs sentinel node biopsy), radiation therapy, anti-HER2 therapy (pertuzumab vs. pyrotinib), chemotherapy (yes vs. no)

CONTACTS AND LOCATIONS:
Overall Officials: Keda Yu, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Keda Yu, Shanghai, China

IPD SHARING:
Plan to Share IPD: No